CLINICAL TRIAL: NCT05607628
Title: Weight Loss Intervention With Lean Muscle Mass Retention (WLMR) Study
Brief Title: Weight Loss Intervention With Lean Muscle Mass Retention
Acronym: WLMR
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Singapore Institute of Food and Biotechnology Innovation (Other Government)
Responsible Party: Principal Investigator, JeyaKumar Henry, Principal Investigator, Singapore Institute of Food and Biotechnology Innovation
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 2022/00205
Record Dates: First submitted 2022-09-22; First posted 2022-11-07 (Actual); Last update posted 2022-11-07 (Actual); Status verified 2022-11

CONDITIONS: Overweight and Obesity
Keywords: Body Weight; Body Fat; Muscle Mass
MeSH Terms: conditions — Overweight; Obesity; Body Weight

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Low-Calorie Control Group (Active Comparator): The control group will receive 2x calorie-restricted balanced meals per day, each consisting of a portion of animal proteins (~20g), a portion of vegetables, and a portion of starch (rice/ noodles) per meal. The group will also receive a mid-morning beverage in the form of a malted drink (~150 kcal and ~5g protein). The third meal of the day and any additional snacks will be left to the free choice of the participants, with calorie advice provided by study dietitian. Calorie restriction aims to reduce body weight of individual participants by ~5 - 10%.
  The group will also be asked to undergo a supervised mixed exercise regime three days per week, 1 hour per day. The mixed exercise regime will consist of 2 sessions of resistance training and 1 session of aerobic training.
  Interventions: Combination Product: Low Calorie Animal Protein Meals
- Low-Calorie Treatment Group (Active Comparator): The treatment group will receive 2x calorie-restricted balanced meals per day, each consisting of a portion of plant proteins (~25g), a portion of vegetables, and a portion of starch (rice/noodles) per meal. The group will also receive a mid-morning beverage, in the form of a soy-based, plant protein beverage (~120 kcal and 13g protein). The third meal of the day and any additional snacks will be left to the free choice of the participants, with calorie advice provided by study dietitian. Calorie restriction aims to reduce body weight of participants by ~5 - 10%.
  The group will also be asked to undergo a supervised mixed exercise regime three days per week, 1 hour per day. The mixed exercise regime will consist of 2 sessions of resistance training and 1 session of aerobic training.
  Interventions: Combination Product: Low Calorie Plant Protein Meals

INTERVENTIONS:
Combination Product: Low Calorie Animal Protein Meals — Consume reduced calorie ready meals with animal proteins to substitute participants' two main meals/day plus a serving of malted beverage to be consumed every day for a period of 16 weeks. Additional supervised exercise regime made up of 2 hours of resistance training plus 1 hour of aerobic training per week for a period of 16 weeks.
  Arms: Low-Calorie Control Group
Combination Product: Low Calorie Plant Protein Meals — Consume reduced calorie ready meals with plant proteins to substitute participants' two main meals/day plus a serving of soy-based plant protein beverage to be consumed every day for a period of 16 weeks. Additional supervised exercise regime made up of 2 hours of resistance training plus 1 hour of aerobic training per week for a period of 16 weeks.
  Arms: Low-Calorie Treatment Group

SUMMARY:
Overweight and obesity (i.e., excess body fat) is a worldwide health problem, which predisposes individuals to various metabolic diseases. Weight loss through lifestyle modifications such as dietary calorie restrictions and/or exercise are effective approaches to reduce excess body fat. However, lean muscle mass loss is often an undesired outcome associated with weight loss, which should be avoided, particularly in older adults, who are also faced with declining anabolic responses to dietary protein intake. Given the increased interest and popularity of plant-based diets, in this study we will compare two distinct calorie-restricted, weight loss diets, both supplemented with weekly exercise, predominantly consisting of either plant-based proteins or animal-based proteins on changes in total body weight, body fat and lean muscle mass, as well as associated changes in metabolic health.

DETAILED DESCRIPTION:
Overweight and obesity is a worldwide health problem which are linked to a plethora of age associated chronic diseases such as diabetes, cardiovascular diseases, hypertension and certain cancers. Lifestyle modifications including calorie-restricted diet and/or exercise are effective, non-invasive strategies to combat this burden. However, due to the age-associated muscle atrophy, consisting of reduced muscle functional status and anabolic resistance, calorie restriction to combat obesity is complicated by concomitant loss of skeletal muscle strength and function. Furthermore, in recent times, due to reasons of sustainability and health, there have been substantial attention on the use of alternative proteins to meet dietary protein requirements.

While increased intake of animal proteins is effective in preserving lean muscle mass, to what extent they apply for plant proteins are still a matter of intense debate. Therefore, in this study we will evaluate and compare two distinct calorie restricted dietary interventions, one predominantly consisting of plant-based proteins and another predominantly consisting of animal-based proteins, both supplemented with increased exercise, on their effectiveness to reduce body fat and preserving lean muscle mass. This will be a 16 week, parallel design, randomized dietary intervention trial, in older Chinese adults, with each volunteer being provided with 2 of their 3 main meals per day, along with a mid-morning beverage, made predominantly of either plant protein or animal protein sources and being asked to undertake 3 hours of additional exercise per week. More details provided in sections below.

ELIGIBILITY:
Inclusion Criteria:

* Male or Female
* Chinese ethnicity
* Age between 40 to 69 years
* Able to give informed consent
* Body Mass Index (BMI) between 23.0 to 32.5 kg/m2

Exclusion Criteria:

* Smoking
* Having allergies or intolerances to any common food ingredients including eggs, fish, milk, peanuts, and tree nuts, shellfish, soya, wheat, gluten, cereal, fruits, dairy products, meat, vegetable, sugar and sweetener, natural food colourings or flavourings, etc
* Following special diets or having intentional dietary restrictions (e.g, vegetarians/vegans)
* Not willing to stop consumption of probiotic or prebiotic supplements within 4 weeks prior to start of study if currently taking these, as well as during study participation
* Not willing to adhere to diet modification as in the study protocol
* Not willing to adhere to the exercise regime as in the study protocol
* Taking part in strenuous physical activities
* Not willing to stop any strenuous activity during or within 24 hours of test days (for those actively participating in sports at the competitive and/or endurance levels)
* Having glucose-6-phosphate dehydrogenase deficiency (G6PD deficiency)
* Having alcohol consumption on > 4 days per week with ≥ 6 alcoholic drinks per week
* Having sustained elevation of blood pressure (>160/95 mm Hg)
* Having previously undergone any gastrointestinal surgery or having history of gastrointestinal disorders
* Having a history of heart, liver, kidney, blood disorders (e.g., thalassemia) or thyroid dysfunctions
* Diabetic
* Having history of tuberculosis, HIV, Hepatitis B or Hepatitis C infections
* Having any prescription medication or any other alternative medicines or supplements which may interfere with study measurements in the in the opinion of the study investigators
* Having antibiotics or suffering from diarrhea within the last 3 months
* Having donated blood within 4 weeks of study participation
* Having poor veins or having history of severe vasovagal syncope (blackouts or fainting) from blood draws
* Having more than 5% weight loss or gain over the past 3 months
* Having metallic implants, pacemaker in the body
* Having claustrophobia
* Having a musculoskeletal injury, joint or peripheral vascular disease sufficient to impede exercise (such as hip arthritis, foot, ankle problems or pain)
* Having severe exercise-induced asthma
* Staff of Wilmar International and/or Singapore Institute of Food and Biotechnology Innovation (SIFBI)
* For female volunteers: menstruation within past 12 months or being on hormone replacement therapy

Ages: 40 Years to 69 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2022-07-18 (Actual); Primary Completion 2022-12-15 (Estimated); Study Completion 2022-12-15 (Estimated)

PRIMARY OUTCOMES:
Body Mass | 16 weeks (from first to final measurement visits)
  kg
Body Fat % | 16 weeks (from first to final measurement visits)
Muscle Mass | 16 weeks (from first to final measurement visits)
  kg

SECONDARY OUTCOMES:
HbA1c | 16 weeks (from first to final measurement visits), measured every 8 weeks
  mmol/mol (%)
Fasting glucose | 16 weeks (from first to final measurement visits), measured every 4 weeks
  mmol/L
Fasting insulin | 16 weeks (from first to final measurement visits), measured every 4 weeks
  pmol/L
Oral glucose tolerance test | 16 weeks (from first to final measurement visits), measured every 8 weeks
  mmol/L
Blood lipid profile (HDL, LDL, Total Cholesterol, Triglyceride) | 16 weeks (from first to final measurement visits), measured every 4 weeks
  mmol/L
C-Reactive Protein | 16 weeks (from first to final measurement visits), measured every 8 weeks
  mg/L
IL-6 (Interleukin 6) | 16 weeks (from first to final measurement visits), measured every 8 weeks
  pg/mL
TNF-α (Tumor Necrosis Factor - alpha) | 16 weeks (from first to final measurement visits), measured every 8 weeks
  pg/mL
Leptin | 16 weeks (from first to final measurement visits), measured every 8 weeks
  ng/mL
β-hydroxybutyrate | 16 weeks (from first to final measurement visits), measured every 8 weeks
  mmol/L
Acetoacetate | 16 weeks (from first to final measurement visits), measured every 8 weeks
  mcg/mL
TMAO (Trimethylamine N-Oxide) | 16 weeks (from first to final measurement visits), measured every 8 weeks
  μM

CONTACTS AND LOCATIONS:
Locations (1):
- Clinical Nutrition Research Centre, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No